CLINICAL TRIAL: NCT03358459
Title: Omics-based Precision Medicine of Epilepsy Being Entrusted by Key Research Project of the Ministry of Science and Technology of China
Brief Title: Omics-based Precision Medicine of Epilepsy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Collaborators: Huashan Hospital (Other); Peking University First Hospital (Other); Peking University People's Hospital (Other); Xiangya Hospital of Central South University (Other); First Affiliated Hospital of Chongqing Medical University (Other); Children's Hospital of Chongqing Medical University (Other); Xuanwu Hospital, Beijing (Other); Capital Medical University (Other); Second Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Yi Wang, vice prsident, Fudan University
Other Study IDs: 2016YFC0904400(1)
Record Dates: First submitted 2017-11-26; First posted 2017-11-30 (Actual); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Epilepsy Idiopathic; Clinical Disease and/or Syndrome; Gene Mutation
Keywords: phenotype; genotype
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — serum 2 ml ; whole blood 3 ml;
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- EP: For diagnosis non-acquired epilepsy;
  Interventions: Other: non

INTERVENTIONS:
Other: non — non

SUMMARY:
Epilepsy is a major disease of the nervous system (WHO, 2015), as well as the second most common neural disease. It has been recorded that there have been 65 million epilepsy patients all over the world, more than 10 million in China, resulted in high morbidity, high mortality, heavy social and social psychological burden. Due to complex etiology, which genetic playing a large part for 70%-80%, easy to recurrent, as well as various seizure types, a great heterogeneity in clinical manifestation, epilepsy is difficult to treat in general, at least 33% patients. At present, It's still a big challenge in early warning, choice of treatment, efficacy and severe adverse reaction rate, prognosis assessment. Lack of precise diagnosis based genetic and molecular bio-markers for treatment are the main key points. Recently, clinical phenotype classifications of epilepsy have been refined, the exist researches had made a progress in gene mutation mechanism and targeted therapy, which pushed epilepsy being another disease could be precise treated after tumor. It's sure to provide a breakthrough for another neural diseases if epilepsy precise treatment project are successful.

DETAILED DESCRIPTION:
Research projects:

Part 1: Based on already existed large samples of epilepsy clinical cases, choose 2,0000 non-acquired epilepsy patients for clinical general phenotype and middle phenotype(EEG and MRI) data collection to further multi-dimensional standardization measure and evaluate. Through metabolic detection to define micro-phenotype. Establish a standardized clinical and biological samples database.

Part 2: By NGS technology to sequence for all cases, including family members, then require genotype. To test brain tissue DNA somatic mutation, which MRI negative and had an operation. To verify the newly discovered pathogenic candidate genes and carry on functional studies. Finally, to draw epileptic genetic mutations mapping in Chinese people.

Part 3: Integrated clinical and genetic epilepsy phenotypic data, combined with neural EEG and image bitmap data points for bio-markers analysis, included early warning, classification of diagnosis, curative effect prediction and epilepsy con-morbidity disease.

ELIGIBILITY:
Inclusion Criteria:

* non-acquired epilepsy; family involved(children, father and mother); Han nationality; Consent and will to follow up

Exclusion Criteria:

* Acquired epilepsy; Very low birth weight infant

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 15000 children and adolescent patients; 5000 adult patients
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2017-11-25 (Actual); Primary Completion 2017-11-26 (Actual); Study Completion 2018-07-01 (Estimated)

PRIMARY OUTCOMES:
The important bio-markers for the efficient therapy and prognosis | 2017.02-2018.07
  the gene mutation or chromosome missing or duplication

CONTACTS AND LOCATIONS:
Overall Officials: Wang yi, Dr, Principal Investigator — leader
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
epilepsy patients with genotype and phenotype can be shared with other collaborators

REFERENCES:
- [Background] EpiPM Consortium. A roadmap for precision medicine in the epilepsies. Lancet Neurol. 2015 Dec;14(12):1219-28. doi: 10.1016/S1474-4422(15)00199-4. Epub 2015 Sep 20. PMID 26416172